CLINICAL TRIAL: NCT03170466
Title: Primary Palliative Care in Heart Failure: A Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Arnold, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PRO16090248; K01HL133466-01 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-05-31 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure
Keywords: Palliative care
MeSH Terms: conditions — Heart Failure | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Palliative Care (Experimental): The intervention will be delivered through four primary mechanisms. First, an existing HF nurse will deliver the intervention to patients during regularly scheduled visits. Second, telephone calls will reinforce topics. Third, patients will regularly report symptoms through the MyUPMC patient portal. Fourth, the nurse will act as a liaison to communicate concerns to the patient's cardiologist and primary care physician, as well as facilitating other resources (e.g., home health). In addition, follow-up assessments will be completed via phone or email at least 2 weeks post-intervention delivery. Caregivers will complete surveys during the first in-person visit and then during the follow-up assessments.
  Interventions: Behavioral: Primary Palliative Care
- Usual Care (No Intervention): Patients randomized to the control arm of this study will continue to receive the standard of high-quality HF care provided to all patients. Control patients may still receive palliative care outside of the study.

INTERVENTIONS:
Behavioral: Primary Palliative Care — The intervention will span 4 domains: symptom management (e.g., dyspnea), psychosocial support (e.g., anxiety), advance care planning (e.g., understanding prognosis and electing a proxy) and care coordination (e.g., communication across providers).
  Other Names: Supportive care
  Arms: Primary Palliative Care

SUMMARY:
Patients with advanced heart failure (HF) typically experience significant burdens that negatively impact their quality of life. Although palliative care has been shown to improve patient outcomes in other serious illnesses, insufficient data exist to support its use in HF. Furthermore, the demand for palliative care in serious illness outstrips the available supply of certified palliative care clinicians. This pilot trial will assess the feasibility and acceptability of training cardiology nurses in basic palliative care skills and their ability to deliver this care alongside usual HF management.

DETAILED DESCRIPTION:
Patients with advanced heart failure (HF) suffer from significant pain, fatigue, difficulty breathing, anxiety, and depression. Palliative Care (PC) is a medical specialty designed to focus on relieving patient suffering by providing an extra layer of support on top of usual care. To date, there has been little research on the impact of PC in HF. We will conduct a randomized clinical trial to assess the feasibility, acceptability, and perceived effectiveness of training cardiology nurses in PC and administering PC to their patients. Patients will be randomized into either the usual care group or the intervention group. Usual care participants will receive their care with no alterations, and intervention participants will receive the PC intervention from their nurse on top of their usual care. Both groups will complete health-related surveys on tablet computers, via email, and/or via telephone. In the intervention group, these answers will be used to tailor the intervention to the specific patient's needs. Caregivers will also be recruited into the study, and will complete surveys similar to the patients via the aforementioned methods.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class III or IV Heart Failure
* 2 or more hospitalizations in the past year due to Heart Failure

Exclusion Criteria:

* Less than 40 years old
* Currently awaiting a transplant
* Received outpatient palliative care within the past 12 months
* Pregnant or intends to be within the next 12 months
* No regular phone access
* Not fluent in English
* Failed the Callahan 6-item Screener
* Does not intent to regularly attend clinic for the next 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling 30 patients via attempting to enroll 30 patients | One year
  We will assess the feasibility of enrolling 30 patients by attempting to enroll 30 patients.

SECONDARY OUTCOMES:
Intervention Acceptability | Two years
  We will evaluate acceptability of the intervention through interviews with patients, caregivers, and healthcare providers.
Intervention Fidelity via the Intervention Fidelity Monitoring Report | Two years
  We will assess intervention fidelity by audio-recording the interventions and having independent reviewers listen to them and complete our Intervention Fidelity Monitoring Report.

CONTACTS AND LOCATIONS:
Overall Officials: Dio Kavalieratos, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Heart Vascular Institute, White Oak, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03170466/ICF_000.pdf